CLINICAL TRIAL: NCT02078466
Title: Assessment of Functional Ability and Follow-up at Home for Older Medical Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: VIA University College (Other); Institute of public health, department of nursing sciences, Århus University, Denmark (Other)
Responsible Party: Principal Investigator, Louise Møldrup Nielsen, PhD student, Occupational Therapist, Aarhus University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Functional ability in older
Record Dates: First submitted 2014-03-01; First posted 2014-03-05 (Estimated); Last update posted 2016-12-12 (Estimated); Status verified 2016-12

CONDITIONS: Geriatric Disorder
Keywords: Functional assessment; readmission; acute care; older medical patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): Usual care
- Assessment of functional ability (Experimental): Assessment of functional ability and follow-up at home
  Interventions: Other: Assessment of functional ability and follow-up at home

INTERVENTIONS:
Other: Assessment of functional ability and follow-up at home — Assessment of functional ability and follow-up at home
  Arms: Assessment of functional ability

SUMMARY:
The aim of this study is to examine the effect of an intervention that consist of assessment of functional ability, rehabilitation plan and follow-up at home for older medical patients.

The hypothesis is that assessment of functional ability, development of rehabilitation plan and follow-up at home reduce the older medical patient's risk of readmission. Also the intervention is expected to reduce mortality, number of contacts to general practitioners and emergency physician

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to Medical Visitations Section (MVA) Aarhus University Hospital
* Aged 65+
* Resident in City of Aarhus

Exclusion Criteria:

* Patients admitted from nursing home
* Patients transferred to other hospital departments
* Patients terminally ill

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 380 (Actual)
Dates: Start 2014-03; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Readmission | Readmission in 26 weeks

SECONDARY OUTCOMES:
Readmission | Readmission in 30 days
Mortality | Mortality in 26 weeks
Number of contacts with GP | 26 weeks
Number of contacts with emergency Physician | 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hans Kirkegaard, Professor, Principal Investigator — Center for Acute Research Aarhus University Hospital
Locations (1):
- Medicinsk Visitationsafsnit, Aarhus, Denmark

REFERENCES:
- [Derived] Nielsen LM, Maribo T, Kirkegaard H, Petersen KS, Lisby M, Oestergaard LG. Effectiveness of the "Elderly Activity Performance Intervention" on elderly patients' discharge from a short-stay unit at the emergency department: a quasi-experimental trial. Clin Interv Aging. 2018 Apr 26;13:737-747. doi: 10.2147/CIA.S162623. eCollection 2018. PMID 29731615